CLINICAL TRIAL: NCT00087958
Title: Phase II Multi-Center, Open-Label, Non-Randomized Study of Intravenous RPR109881 Given Every 3 Weeks in Patients With Metastatic Breast Cancer Progressing After Therapy With Anthracyclines, Taxanes and Capecitabine
Brief Title: Intravenous RPR109881 in Male or Female Patients With Advanced Breast Cancer Who no Longer Respond to Anthracycline, Taxane and Capecitabine Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EFC6088; XRP9881B/2001; EUDRACT : 2004-000572-14
Record Dates: First submitted 2004-07-16; First posted 2004-07-20 (Estimated); Last update posted 2009-05-01 (Estimated); Status verified 2009-04

CONDITIONS: Breast Cancer
Keywords: Metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — larotaxel

INTERVENTIONS:
Drug: XRP9881

SUMMARY:
The purpose of this clinical trial is to determine if the investigational drug is able to reduce/shrink advanced breast cancer tumors in patients who no longer benefit from anthracyclines, taxanes and capecitabine.

DETAILED DESCRIPTION:
All patients in this trial will receive the investigational (chemotherapy) drug at an optimal dose as determined by previous clinical trials. The investigational drug is given through a vein once every three weeks. This drug prevents tumor cells from dividing, so they may stop growing or die.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for this trial you must:

* Have a diagnosis of breast cancer that is now metastatic (meaning the cancer has spread beyond its original location) or a recurrence of the cancer in its original location that cannot be removed by surgery.
* Have received previous treatment with anthracyclines (e.g. doxorubicin [Adriamycin or Doxil] or epirubicin [Ellence]), taxanes (paclitaxel [Taxol or Abraxane] or docetaxel [Taxotere]) and capecitabine (e.g. Xeloda) for your breast cancer and your doctor has determined that these treatments are no longer of benefit to you.
* Be at least 18 years of age
* Not be taking other treatments for your cancer at the time you enter the trial.
* Not be pregnant
* Additionally, there are other criteria for study entry that a doctor participating in this study will need to review in detail with you and clinical assessments may need to be performed (lab tests, CT scans).

Exclusion Criteria:

* None listed here. Can be discussed with your doctor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2004-08; Primary Completion 2007-02 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Objective response rate as assessed by Response Evaluation Criteria in Solid Tumors

SECONDARY OUTCOMES:
Progression free survival, overall survival, composite event of CR, PR and stable disease > or = to 12 weeks
Time to tumor response and duration of response.
Safety analyses based on incidence, severity, chronicity and cumulative nature of TEAEs.

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (15):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Bogotá, Colombia
- Sanofi-Aventis Administrative Office, Hørsholm, Denmark
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Midrand, South Africa
- Sanofi-Aventis Administrative Office, Seoul, South Korea
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Geneva, Switzerland
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)